CLINICAL TRIAL: NCT04740151
Title: Individualized vs Standard PEEP in Thoracic Surgery: Effects on Respiratory Mechanics and Intra- and Postoperative Oxygenation
Brief Title: Individualized PEEP in Thoracic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Trieste (Other)
Responsible Party: Principal Investigator, Lucia Comuzzi, Principal Investigator, University of Trieste
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 49/2017
Record Dates: First submitted 2021-01-15; First posted 2021-02-05 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Thoracic Surgery; One-lung Ventilation; Respiratory Mechanics; Artificial Respiration
Keywords: Individualized PEEP; One-lung ventilation; Oxygenation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BEST PEEP (Experimental): During OLV an individualized PEEP will be applied i.e. the one corresponding to the lower driving pressure, + 2 cmH2O
  Interventions: Procedure: Best PEEP
- STANDARD PEEP (Active Comparator): During OLV a PEEP of 5 cmH2O will be applied
  Interventions: Procedure: Standard PEEP

INTERVENTIONS:
Procedure: Best PEEP — In OLV, the investigator will perform a PEEP decremental titration trial, decreasing PEEP from 16 to 4 cmH2O (steps of 2-cmH2O, lasting 1 minute). At the end of every step driving pressure (Pplat-PEEP) will be calculated, and the PEEP corresponding to the lowest driving pressure + 2cmH2O will be set.
  Arms: BEST PEEP
Procedure: Standard PEEP — In OLV, a PEEP of 5 cm H2O will be set.
  Arms: STANDARD PEEP

SUMMARY:
Intraoperative protective ventilation with low tidal volumes (TV), positive end-expiratory pressure (PEEP) and possibly lung recruitment maneuvers (RMs) reduces postoperative pulmonary complications. In thoracic surgery, in one-lung ventilation (OLV), the evidence is lacking. However, in this context protective ventilation with PEEP titration is related to better intraoperative oxygenation and respiratory mechanics. It is not clear whether this strategy is associated also with better postoperative oxygenation and less postoperative pulmonary complications.

DETAILED DESCRIPTION:
In this randomized controlled trial the investigators will enroll 42 patients scheduled for elective thoracic surgery (minithoracotomic or video-assisted thoracoscopic segmentectomies and lobectomies). Patients will be randomized in two groups: BEST PEEP and STANDARD PEEP. In OLV the investigator will set a TV = 5ml/kg IBW in volume control ventilation (VCV) and an adequate respiratory rate (RR) to keep PaCO2 < 60 mmHg. With the patient in lateral decubitus and open chest, a cycling step RM (in pressure control ventilation, RR =10/min, I:E=1:1, up to Paw = 40 cmH20 with a PEEP = 20 cmH2O, lasting 2.5 minutes) and a PEEP decremental titration trial (in VCV, from 16 to 4 cmH2O) will be performed to all patients. Then, after another RM, in STANDARD PEEP group a PEEP of 5 cmH2O will be set, and in BEST PEEP group an individualized PEEP (the one corresponding to the lower driving pressure, +2 cmH2O) will be applied till the end of surgery. A blood gas analysis will be performed before surgery, with the patient in supine position breathing room air (T1). The respiratory mechanics (Ppeak, Pplateau, PEEP, driving pressure) and blood gas (PaO2, PaCO2, pH, HCO3, lactates) parameters will be then collected at the following time points: T2 - 5 minutes after induction, patient supine, two lung ventilation; T3 - lateral decubitus, chest open, OLV, before RM; T4 - 10 minutes after second RM; T5, 6, 7 - every hour after T4; T8 - at the end of OLV, before lung re-expansion; T9 - patient supine, two lung ventilation, before neuromuscular block reversal. Postoperatively all patients will spend at least one hour in a Recovery Room, in oxygen-therapy through a Venturi mask with FiO2 = 60%. A blood gas analysis and data about pain (NRS scale 0-10) and sedation (Ramsey score) will be collected at 1 hour postoperatively (T10). The primary outcome of the study is intra- and postoperative oxygenation and secondary outcomes are intraoperative respiratory mechanics parameters.

ELIGIBILITY:
Inclusion criteria:

* Patient's consent to the trial
* Candidate to elective lung lobectomy or segmentectomy (minimally invasive thoracotomy or video-assisted thoracoscopy)
* ASA class 1-3
* BMI < 30 kg/m2

Exclusion criteria:

* Pregnancy
* Previous pneumothorax,
* Emphysematous bullae
* Severe COPD
* METs < 4 due to cardiac disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-01-04 (Actual); Primary Completion 2021-12-04 (Actual); Study Completion 2021-12-05 (Actual)

PRIMARY OUTCOMES:
Change of oxygenation | The blood gas analysis will be performed at the time points from T1 to T10 (preoperative, during surgery and 1 hour postoperative). The investigators will perform intra- and inter-group comparisons.
  Oxygen arterial partial pressure/fraction of inspired oxygen (PaO2/FiO2)

SECONDARY OUTCOMES:
Change of driving pressure | The respiratory mechanics parameters will be collected at the time points from T2 to T9 (during surgery). The investigators will perform intra- and inter-group comparisons.
  Driving pressure = Pplateau -PEEP
Change of plateau pressure | The respiratory mechanics parameters will be collected at the time points from T2 to T9 (during surgery). The investigators will perform intra- and inter-group comparisons.
  Airway pressure during an end-inspiratory pause
Change of static respiratory system compliance | The respiratory mechanics parameters will be collected at the time points from T2 to T9 (during surgery). The investigators will perform intra- and inter-group comparisons.
  Cstat = TV/(Pplat-PEEP)
Change of respiratory rate | The parameter will be collected at the time points from T2 to T9 (during surgery). The investigators will perform intra- and inter-group comparisons.
  Respiratory rate set on the ventilator
Change of carbon dioxide | The blood gas analysis will be performed at the time points from T1 to T10 (preoperative, during surgery and 1 hour postoperative). The investigators will perform intra- and inter-group comparisons.
  Carbon dioxide arterial partial pressure
Change of end expiratory carbon dioxide partial pressure | The respiratory parameters will be collected at the time points from T2 to T9 (during surgery). The investigators will perform intra- and inter-group comparisons.
  Carbon dioxide end-expiratory partial pressure
Change of pH | The blood gas analysis will be performed at the time points from T1 to T10 (preoperative, during surgery and 1 hour postoperative). The investigators will perform intra- and inter-group comparisons.
  Arterial pH
Lactate | The blood gas analysis will be performed at the time points from T1 to T10 (preoperative, during surgery and 1 hour postoperative). The investigators will perform intra- and inter-group comparisons.
  Arterial lactate

CONTACTS AND LOCATIONS:
Overall Officials: Lucia Comuzzi, Principal Investigator — Azienda Sanitaria Universitaria Giuliano Isontina (ASU GI)
Locations (1):
- Azienda Sanitaria Universitaria Giuliano-Isontina, Cattinara Hospital, Trieste, Italy

IPD SHARING:
Plan to Share IPD: No